CLINICAL TRIAL: NCT03468582
Title: Pilot Study Using 123I Radiolabeled 3BNC117 SPECT/CT to Image HIV Reservoir in Chronically Infected HIV Patients
Brief Title: 123I Radiolabeled 3BNC117
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, John O. Prior, Head of nuclear medicine and molecular imaging department, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-01003
Record Dates: First submitted 2018-02-12; First posted 2018-03-16 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Monocentric, open-label and uncontrolled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 123I radiolabeled 3BNC117 (Experimental): 123I radiolabeled 3BNC117
  Interventions: Combination Product: 123I radiolabeled 3BNC117

INTERVENTIONS:
Combination Product: 123I radiolabeled 3BNC117 — 123I radiolabeled 3BNC117

SUMMARY:
The conventional way to control HIV infection is the usage of a drug cocktail capable of suppressing the viral replication cycle, commonly known as antiretroviral therapy (ART). Despite effective ART it is not possible to eradicate HIV. The virus hides in particular cells to form the latent HIV-reservoir.[1-9] Studies that emphasise on revealing hidden reservoirs would aid in designing novel therapeutic strategies for controlling HIV infection. Molecular imaging by SPECT/CT has the potential to reveal hidden reservoirs of HIV virus that are not eliminated by currently used drugs capable of suppressing and thereby controlling the viral replication cycle in HIV infected patients. New approaches, necessary to prevent and treat HIV-1 infection, are gradually emerging. A new generation of highly potent broadly neutralizing antibodies (bN/Abs) may represent a promising approach to combating HIV-1 infection.[10] The broadly neutralizing antibody 3BNC117 antibody that can mimic human CD4 binding targeted against the HIV gp120 envelope protein has been tested in various clinical trials.[11-14] It has found to be safe and effective in reducing viraemia and to improve host humoral responses in HIV-1 infected individuals, and to have effect on viral rebound in patients who are kept off antiretroviral treatment briefly for experimental purpose.

Imaging of simian immunodeficiency virus (SIV) infection by PET/CT has been successfully performed in nonhuman primates with a 64Cu-labeled SIV gp120-specific antibody called 7D3.[15] This study aims to use a similar approach in human with the 3BNC117 antibody. The 3BNC117 antibody has been successfully radiolabeled with iodine 123. The half-life of this radioisotope is appropriate for antibody imaging in nuclear medicine. Radiolabeled 123I 3BNC117 was shown to keep a good immunoreactivity for gp120. By using state of the art SPECT scanner a semi-quantitative image will be obtained. In addition, the absence of any chelator and the well known use of iodine-123 in clinic make it suitable for human intervention.

No HIV imaging in human has been achieved yet, which is however fundamental to understand some key steps in the pathogenesis of HIV-induced immunodeficiency. This research opens promising opportunities for drug and vaccine development. Indeed, identification of virus reservoirs in treated patients would facilitate the development of strategies for eradicating these reservoirs or for extending latency period.

DETAILED DESCRIPTION:
The conventional way to control HIV infection is by use of a cocktail of drugs capable of suppressing the viral replication cycle, commonly known as antiretroviral therapy (ART). Despite effective ART it is not possible to eradicate HIV. The virus hides in particular cells to form the latent HIV-reservoir and antiviral agents have no effect on these latently infected HIV cells.[1-9] Studies by Chomont et al. identified particular CD4 T cell subsets that serve as key cellular compartment for latent HIV-1 reservoir in blood.[6] A later study has identified memory CD4 T cells with stem-cell like properties as a minor latent HIV-1 reservoir.[7] A major part of this reservoir is in the lymphoid tissue which constitute the predominant site for lymphocytes. One recent study has identified follicular T helper cells (TFH) of lymph nodes as major CD4 T cell compartments for HIV-1 replication, production and infection.[8] Further characterisation of the different CD4 T cell population has identified a specific cell population expressing PD-1(+) as the major CD4 T cell compartment in blood and lymph nodes for production of replication competent and infectious HIV-1.[9] Thus, studies that emphasise on revealing hidden reservoirs would aid in designing novel therapeutic strategies for controlling HIV infection. Molecular imaging by SPECT/CT has the potential to reveal hidden reservoirs of HIV virus that are not eliminated by use of currently used drugs capable of suppressing and thereby controlling the viral replication cycle in HIV infected patients.

As discussed above, even though ART can suppress virus replication and can limit disease progression, it fails to eradicate the virus, and suppression requires lifelong therapy, which may have side effects and poses a risk of the development of resistance. New approaches necessary to prevent and treat HIV-1 infection in order to restrict the epidemic and to strengthen nascent efforts in finding a cure are gradually emerging. A new generation of highly potent broadly neutralizing antibodies (bNAbs) may represent a promising approach to combating HIV-1 infection.[10] Many sites on the viral envelope can be recognized by bNAbs.

The broadly neutralising antibody 3BNC117 directed against the HIV gp120 envelope protein, can mimic human CD4 binding and can neutralize 195 out of 237 HIV-1 strains.[11] The first human phase I dose escalation study using 3BNC117, has shown to be safe and effective in transiently reducing viraemia in chronic HIV-1 infected individuals.[12] A subsequent study (ClinicalTrial.gov identifier:NCT02018510) demonstrated improved host humoral immune response in infected individuals treated with 3BNC117 antibody as compared to untreated individuals.[13] Furthermore, a phase IIa open labelled trial by the same group of researchers at Rockefeller University, NY has been carried out to evaluate the capacity of this antibody to suppress viral rebound in infected individuals during a brief treatment interruption of anti-retroviral therapy.[14] Another such trial is currently ongoing (ClinicalTrial.gov identifier: NCT02446847).

Imaging of simian immunodeficiency virus (SIV) infection by PET/CT has been successfully performed in nonhuman primates with a 64Cu-labeled SIV gp120-specific antibody called 7D3.[15] This study aims to use a similar approach in human with the 3BNC117 antibody. The 3BNC117 antibody has been successfully radiolabeled with iodine-123. The half-life of this radioisotope is appropriate for antibody imaging in nuclear medicine. Radiolabeled 123I-3BNC117 was shown to keep a good immunoreactivity in vitro for gp120. By using state of the art SPECT scanner a semi-quantitative image will be obtained. In addition, the well known use of iodine-123 in clinic and the absence of chelator makes it suitable for human intervention.

No HIV imaging in human has yet been achieved, which is however fundamental to understand some key steps in the pathogenesis of the HIV-induced immunodeficiency. This research opens promising opportunities for monitoring the size of the HIV reservoir and for drug and vaccine development. Indeed, identification of virus reservoirs in treated patients would facilitate the development of strategies for eradicating these reservoirs or for extending latency period.

ELIGIBILITY:
Inclusion Criteria:

* Subject newly diagnosed with HIV in a chronic phase requiring the introduction of an antiretroviral treatment (ART)
* Age 18 to 55
* HIV-1 infection confirmed by ELISA and immunoblot
* Plasma HIV-1 RN/A > 5000 copies/ml
* Current CD4 cell count > 200 cells/μl
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Primary infected HIV
* Currently on ART
* Participation in another clinical study of an investigational product currently or within past 30 days
* Pregnancy or lactation;
* History of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months;
* Patient report, or chart history, of significant coronary artery disease, myocardial infarction, percutaneous coronary intervention with placement of cardiac stents;
* Uncontrolled hypertension, as defined by a systolic blood pressure > 180 and/or diastolic blood pressure > 120, in the presence or absence of anti-hypertensive medications;
* Any other clinically significant acute or chronic medical condition, such as autoimmune diseases, that in the opinion of the investigator would preclude participation;
* Laboratory abnormalities in the parameters listed below:
* Absolute neutrophil count ≤1 G/l
* Hemoglobin ≤ 10 gm/dL
* Platelet count ≤125 G/l
* ALT ≥ 2.0 x ULN
* AST ≥ 2.0 x ULN
* Total bilirubin ≥ 1.5 ULN
* Creatinine ≥ 1.1 x ULN
* Coagulation parameters ≥ 1.5 x ULN

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Absorbed dose per Organ mGy/MBq | 3 month
  Absorbed dose in the organs at risk is calculated from planar images after organ contouring using OLINDA / EXM software; additionally blood samples (2 mL) is taken before each gamma camera scan to estimate the dose to bone marrow. The blood samples are needed to derive the radiation dose exposure to the bone marrow through the measure of the count rate in the blood sample using a calibrated gamma counter. MIRD (medical internal radiation dosimetry) based methods will provide the contribution to the bone marrow radiation exposure from activity present into the blood.[19] No other additional analysis will be performed on these blood samples.

SECONDARY OUTCOMES:
total number of lesions | 3 month
  Accumulation of 123I-3BNC117 in target organs and HIV reservoirs is delineated in the patients before and after ART treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pantaleo, MD, PhD, Study Director — University of Lausanne Hospitals
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Data will not be shared with third parties having lower protection standards then Switzerland.

REFERENCES:
- [Background] Chun TW, Stuyver L, Mizell SB, Ehler LA, Mican JA, Baseler M, Lloyd AL, Nowak MA, Fauci AS. Presence of an inducible HIV-1 latent reservoir during highly active antiretroviral therapy. Proc Natl Acad Sci U S A. 1997 Nov 25;94(24):13193-7. doi: 10.1073/pnas.94.24.13193. PMID 9371822
- [Background] Chun TW, Carruth L, Finzi D, Shen X, DiGiuseppe JA, Taylor H, Hermankova M, Chadwick K, Margolick J, Quinn TC, Kuo YH, Brookmeyer R, Zeiger MA, Barditch-Crovo P, Siliciano RF. Quantification of latent tissue reservoirs and total body viral load in HIV-1 infection. Nature. 1997 May 8;387(6629):183-8. doi: 10.1038/387183a0. PMID 9144289
- [Background] Finzi D, Hermankova M, Pierson T, Carruth LM, Buck C, Chaisson RE, Quinn TC, Chadwick K, Margolick J, Brookmeyer R, Gallant J, Markowitz M, Ho DD, Richman DD, Siliciano RF. Identification of a reservoir for HIV-1 in patients on highly active antiretroviral therapy. Science. 1997 Nov 14;278(5341):1295-300. doi: 10.1126/science.278.5341.1295. PMID 9360927
- [Background] Wong JK, Hezareh M, Gunthard HF, Havlir DV, Ignacio CC, Spina CA, Richman DD. Recovery of replication-competent HIV despite prolonged suppression of plasma viremia. Science. 1997 Nov 14;278(5341):1291-5. doi: 10.1126/science.278.5341.1291. PMID 9360926
- [Background] Siliciano JD, Kajdas J, Finzi D, Quinn TC, Chadwick K, Margolick JB, Kovacs C, Gange SJ, Siliciano RF. Long-term follow-up studies confirm the stability of the latent reservoir for HIV-1 in resting CD4+ T cells. Nat Med. 2003 Jun;9(6):727-8. doi: 10.1038/nm880. Epub 2003 May 18. PMID 12754504
- [Background] Chomont N, El-Far M, Ancuta P, Trautmann L, Procopio FA, Yassine-Diab B, Boucher G, Boulassel MR, Ghattas G, Brenchley JM, Schacker TW, Hill BJ, Douek DC, Routy JP, Haddad EK, Sekaly RP. HIV reservoir size and persistence are driven by T cell survival and homeostatic proliferation. Nat Med. 2009 Aug;15(8):893-900. doi: 10.1038/nm.1972. Epub 2009 Jun 21. PMID 19543283
- [Background] Buzon MJ, Sun H, Li C, Shaw A, Seiss K, Ouyang Z, Martin-Gayo E, Leng J, Henrich TJ, Li JZ, Pereyra F, Zurakowski R, Walker BD, Rosenberg ES, Yu XG, Lichterfeld M. HIV-1 persistence in CD4+ T cells with stem cell-like properties. Nat Med. 2014 Feb;20(2):139-42. doi: 10.1038/nm.3445. Epub 2014 Jan 12. PMID 24412925
- [Background] Perreau M, Savoye AL, De Crignis E, Corpataux JM, Cubas R, Haddad EK, De Leval L, Graziosi C, Pantaleo G. Follicular helper T cells serve as the major CD4 T cell compartment for HIV-1 infection, replication, and production. J Exp Med. 2013 Jan 14;210(1):143-56. doi: 10.1084/jem.20121932. Epub 2012 Dec 17. PMID 23254284
- [Background] Banga R, Procopio FA, Noto A, Pollakis G, Cavassini M, Ohmiti K, Corpataux JM, de Leval L, Pantaleo G, Perreau M. PD-1(+) and follicular helper T cells are responsible for persistent HIV-1 transcription in treated aviremic individuals. Nat Med. 2016 Jul;22(7):754-61. doi: 10.1038/nm.4113. Epub 2016 May 30. PMID 27239760
- [Background] Klein F, Mouquet H, Dosenovic P, Scheid JF, Scharf L, Nussenzweig MC. Antibodies in HIV-1 vaccine development and therapy. Science. 2013 Sep 13;341(6151):1199-204. doi: 10.1126/science.1241144. PMID 24031012
- [Background] Scheid JF, Mouquet H, Ueberheide B, Diskin R, Klein F, Oliveira TY, Pietzsch J, Fenyo D, Abadir A, Velinzon K, Hurley A, Myung S, Boulad F, Poignard P, Burton DR, Pereyra F, Ho DD, Walker BD, Seaman MS, Bjorkman PJ, Chait BT, Nussenzweig MC. Sequence and structural convergence of broad and potent HIV antibodies that mimic CD4 binding. Science. 2011 Sep 16;333(6049):1633-7. doi: 10.1126/science.1207227. Epub 2011 Jul 14. PMID 21764753
- [Background] Caskey M, Klein F, Lorenzi JC, Seaman MS, West AP Jr, Buckley N, Kremer G, Nogueira L, Braunschweig M, Scheid JF, Horwitz JA, Shimeliovich I, Ben-Avraham S, Witmer-Pack M, Platten M, Lehmann C, Burke LA, Hawthorne T, Gorelick RJ, Walker BD, Keler T, Gulick RM, Fatkenheuer G, Schlesinger SJ, Nussenzweig MC. Viraemia suppressed in HIV-1-infected humans by broadly neutralizing antibody 3BNC117. Nature. 2015 Jun 25;522(7557):487-91. doi: 10.1038/nature14411. Epub 2015 Apr 8. PMID 25855300
- [Background] Schoofs T, Klein F, Braunschweig M, Kreider EF, Feldmann A, Nogueira L, Oliveira T, Lorenzi JC, Parrish EH, Learn GH, West AP Jr, Bjorkman PJ, Schlesinger SJ, Seaman MS, Czartoski J, McElrath MJ, Pfeifer N, Hahn BH, Caskey M, Nussenzweig MC. HIV-1 therapy with monoclonal antibody 3BNC117 elicits host immune responses against HIV-1. Science. 2016 May 20;352(6288):997-1001. doi: 10.1126/science.aaf0972. Epub 2016 May 5. PMID 27199429
- [Background] Scheid JF, Horwitz JA, Bar-On Y, Kreider EF, Lu CL, Lorenzi JC, Feldmann A, Braunschweig M, Nogueira L, Oliveira T, Shimeliovich I, Patel R, Burke L, Cohen YZ, Hadrigan S, Settler A, Witmer-Pack M, West AP Jr, Juelg B, Keler T, Hawthorne T, Zingman B, Gulick RM, Pfeifer N, Learn GH, Seaman MS, Bjorkman PJ, Klein F, Schlesinger SJ, Walker BD, Hahn BH, Nussenzweig MC, Caskey M. HIV-1 antibody 3BNC117 suppresses viral rebound in humans during treatment interruption. Nature. 2016 Jul 28;535(7613):556-60. doi: 10.1038/nature18929. Epub 2016 Jun 22. PMID 27338952
- [Background] Santangelo PJ, Rogers KA, Zurla C, Blanchard EL, Gumber S, Strait K, Connor-Stroud F, Schuster DM, Amancha PK, Hong JJ, Byrareddy SN, Hoxie JA, Vidakovic B, Ansari AA, Hunter E, Villinger F. Whole-body immunoPET reveals active SIV dynamics in viremic and antiretroviral therapy-treated macaques. Nat Methods. 2015 May;12(5):427-32. doi: 10.1038/nmeth.3320. Epub 2015 Mar 9. PMID 25751144
- [Background] Falkowska E, Ramos A, Feng Y, Zhou T, Moquin S, Walker LM, Wu X, Seaman MS, Wrin T, Kwong PD, Wyatt RT, Mascola JR, Poignard P, Burton DR. PGV04, an HIV-1 gp120 CD4 binding site antibody, is broad and potent in neutralization but does not induce conformational changes characteristic of CD4. J Virol. 2012 Apr;86(8):4394-403. doi: 10.1128/JVI.06973-11. Epub 2012 Feb 15. PMID 22345481
- [Background] Shingai M, Nishimura Y, Klein F, Mouquet H, Donau OK, Plishka R, Buckler-White A, Seaman M, Piatak M Jr, Lifson JD, Dimitrov DS, Nussenzweig MC, Martin MA. Antibody-mediated immunotherapy of macaques chronically infected with SHIV suppresses viraemia. Nature. 2013 Nov 14;503(7475):277-80. doi: 10.1038/nature12746. Epub 2013 Oct 30. PMID 24172896
- [Background] Aroua A, Samara ET, Bochud FO, Meuli R, Verdun FR. Exposure of the Swiss population to computed tomography. BMC Med Imaging. 2013 Jul 30;13:22. doi: 10.1186/1471-2342-13-22. PMID 23895057
- [Background] Hindorf C, Glatting G, Chiesa C, Linden O, Flux G; EANM Dosimetry Committee. EANM Dosimetry Committee guidelines for bone marrow and whole-body dosimetry. Eur J Nucl Med Mol Imaging. 2010 Jun;37(6):1238-50. doi: 10.1007/s00259-010-1422-4. PMID 20411259